CLINICAL TRIAL: NCT05990647
Title: Incisional Hernia Impact on Muscular and Postural Function
Brief Title: Impact Evaluation of Incisional Hernia on Muscular and Postural Function
Acronym: IHMPF-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov (Other)
Collaborators: Tashkent state dental institute (Unknown); I.M. Sechenov First Moscow State Medical University (Other); Pirogov Russian National Research Medical University (Other)
Responsible Party: Principal Investigator, Nikita A. Demin, Principal investigator, Republican Specialized Scientific and Practical Medical Center of Surgery Named After V. Vakhidov
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: "EC" №1-2022
Record Dates: First submitted 2023-07-22; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Incisional Hernia
Keywords: incisional hernia; tension dynamometry; raster photostereography; postural balance; hernia repair; bridging technique; Rives-Stoppa; TAR
MeSH Terms: conditions — Incisional Hernia | interventions — Postural Balance

STUDY DESIGN:
Intervention Model Description: Cohort study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Active Comparator): 32 patients who underwent classic abdominal wall anterior components separation and bridged hernia repair.
  Interventions: Diagnostic Test: Dynamometric tension assessment; Diagnostic Test: Postural balance; Diagnostic Test: Assessment of the hernia defect size; Diagnostic Test: Physical activity of patients
- Group II (Active Comparator): 34 patients who underwent posterior components separation with the internal oblique myofascial release by Rives-Stoppa
  Interventions: Diagnostic Test: Dynamometric tension assessment; Diagnostic Test: Postural balance; Diagnostic Test: Assessment of the hernia defect size; Diagnostic Test: Physical activity of patients
- Group III (Active Comparator): 29 patients who underwent posterior components separation with transversus abdominis release (TAR).
  Interventions: Diagnostic Test: Dynamometric tension assessment; Diagnostic Test: Postural balance; Diagnostic Test: Assessment of the hernia defect size; Diagnostic Test: Physical activity of patients

INTERVENTIONS:
Diagnostic Test: Dynamometric tension assessment — Tension dynamometry was carried out using the "Back-Check 600" diagnostic complex by Dr.WOLFF® (GmbH, Germany). The dynamometric stress assessment included tasks for flexion and extension of the body. The functional assessment of the abdominal wall muscles was assessed when preparing the patient for surgery (1-10 days before AWR-abdominal wall reconstruction) and 6 months after AWR.
  Other Names: DT
Diagnostic Test: Postural balance — Postural balance was assessed using raster photostereography and baropodometry on the "DIERS" diagnostic complex by Formetric-4D (GmbH, Germany). When analyzing the topography of the optical field, muscle imbalance is revealed in the form of lateral deviation and inclination of the trunk and pelvis, as well as the values of the angle of kyphosis and lordosis. When conducting baropodometry, the level of displacement of the pressure area on the feet of patients in a static and dynamic position was assessed. Diagnosis of postural balance in patients with incisional ventral hernia was performed a few days before surgical treatment and 6 months after AWR.
  Other Names: PB
Diagnostic Test: Assessment of the hernia defect size — Parameters of the hernial defect, including the volume of the hernial sac, the diameter of the hernial orifice, the ratio of hernia volume to the abdominal cavity volume, were performed using preoperative (1-10 days before AWR) multispiral computed tomography on a GE "BrightSpeed 16" tomograph (General Electric©, USA)
Diagnostic Test: Physical activity of patients — To analyze the physical activity of patients, the measurement of the number of steps was used. The measurements of steps and the amount of distance traveled were carried out using a physical activity monitor - a fitness bracelet "MiBAND" (China). Measurements were taken 10 days before AWR and within 6 months after AWR.
  Other Names: PAP

SUMMARY:
Purpose of study is to assess perioperative functional parameters of the anterior abdominal wall muscles and postural control status in patients with large and giant incisional hernias in a controlled diagnostic study.

The study involved 95 patients (100% completed) with a large or giant incisional hernia of the anterior abdominal wall. The participants were divided into three groups by type of hernia repair: bridged hernia repair, Rives-Stoppa procedure, or TAR technique. Perioperative functional parameters of the anterior abdominal wall muscles were assessed by tension dynamometry. The postural balance assessments were made by raster photostereography.

ELIGIBILITY:
Inclusion Criteria:

* big and giant incisional hernia
* hernia without recurrence
* age 18-75

Exclusion Criteria:

* acute infection diseases
* cancer
* orthopedic diseases
* terminal status
* BMI>39,9

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1-2 weeks before surgical treatment and 6 months after reconstructive hernioplasty of postoperative ventral hernia
  Sensitivity and specificity

CONTACTS AND LOCATIONS:
Overall Officials: Otabek J. Eshonkhodjaev, MD, PhD, Study Chair — Republican specialiazed scientific practical medical center of surgery named after V.V. Vakhidov
Locations (1):
- Republican specialized scientific practical medical center of surgery named after V.V. Vakhidov, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR